CLINICAL TRIAL: NCT02654054
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Elagolix in Combination With Estradiol/Norethindrone Acetate for the Management of Heavy Menstrual Bleeding Associated With Uterine Fibroids in Premenopausal Women
Brief Title: Efficacy and Safety of Elagolix in Combination With Estradiol/Norethindrone Acetate for the Management of Heavy Menstrual Bleeding Associated With Uterine Fibroids in Premenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M12-815
Record Dates: First submitted 2016-01-08; First posted 2016-01-13 (Estimated); Results first posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Uterine Fibroids; Heavy Menstrual Bleeding
Keywords: Elagolix; Elagolix Sodium; Heavy Uterine Bleeding; Heavy Menstrual Bleeding; Leiomyomata; Menorrhagia; ABT-620; Elagolix + E2/NETA; Elagolix + Norethindrone Acetate; HMB
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — elagolix; Estradiol; Norethindrone Acetate; estradiol, norethindrone drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo for both elagolix twice daily (BID) and norethindrone acetate (E2/NETA) once daily (QD)
  Interventions: Drug: Placebo for Estradiol/Norethindrone Acetate; Drug: Placebo for Elagolix
- Elagolix (Experimental): Elagolix 300 mg BID and placebo for E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) QD
  Interventions: Drug: Elagolix; Drug: Placebo for Estradiol/Norethindrone Acetate
- Elagolix + E2/NETA (Experimental): Elagolix 300 mg BID and E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) QD
  Interventions: Drug: Elagolix; Drug: Estradiol/Norethindrone Acetate

INTERVENTIONS:
Drug: Elagolix — Film-coated tablets
  Other Names: ABT-620; elagolix sodium
  Arms: Elagolix; Elagolix + E2/NETA
Drug: Placebo for Estradiol/Norethindrone Acetate — Placebo capsules
  Arms: Elagolix; Placebo
Drug: Estradiol/Norethindrone Acetate — Commercially-available E2/NETA tablets were over-encapsulated to maintain study blinding.
  Other Names: E2/NETA
  Arms: Elagolix + E2/NETA
Drug: Placebo for Elagolix — Film-coated placebo tablets
  Arms: Placebo

SUMMARY:
This study seeks to evaluate the efficacy, safety and tolerability of elagolix alone and in combination with estradiol/norethindrone acetate for the management of heavy menstrual bleeding associated with uterine fibroids in premenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a premenopausal female at the time of Screening.
* Subject has a diagnosis of uterine fibroids documented by a pelvic ultrasound (transabdominal ultrasound/transvaginal ultrasound).
* Subject has heavy menstrual bleeding associated with uterine fibroids as evidenced by menstrual blood loss > 80 mL during each of two screening menses as measured by the alkaline hematin method.
* Subject has negative urine and/or serum pregnancy test in Screening and just prior to first dose.
* Subject has an adequate endometrial biopsy performed during Screening, the results of which show no clinically significant endometrial pathology.

Exclusion Criteria:

* Subject has screening pelvic ultrasound or saline infusion sonohysterography results that show a clinically significant gynecological disorder.
* Subject has history of osteoporosis or other metabolic bone disease.
* Subject has clinically significant abnormalities in clinical chemistry, hematology, or urinalysis.
* Subject has a history of major depression or post-traumatic stress disorder (PTSD) within 2 years of screening, OR a history of other major psychiatric disorder at any time (e.g., schizophrenia, bipolar disorder).
* Subject is using any systemic corticosteroids for over 14 days within 3 months prior to Screening or is likely to require treatment with systemic corticosteroids during the course of the study. Over the counter and prescription topical, inhaled, intranasal or injectable (for occasional use) corticosteroids are allowed.

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 413 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (96):
- United States (92):
  - Summers, Birmingham, AL /ID# 139684, Birmingham, Alabama
  - University of South Alabama /ID# 148763, Mobile, Alabama
  - WCCT Global, LLC /ID# 145666, Costa Mesa, California
  - American Clinical Trials /ID# 147374, Hawaiian Gardens, California
  - Grossmont Ctr Clin Research /ID# 144011, La Mesa, California
  - Long Beach Clinical Trial Serv /ID# 152424, Long Beach, California
  - National Research Institute /ID# 151629, Los Angeles, California
  - University of California, Los Angeles /ID# 144107, Los Angeles, California
  - Beach OBGYN Medical Group /ID# 151414, Newport Beach, California
  - Advanced RX Clinical Research /ID# 149168, Westminster, California
  - Bluebird Clinical Trials, LLC /ID# 144843, Colorado Springs, Colorado
  - Advanced Women's Health Institution /ID# 144108, Greenwood Village, Colorado
  - Medstar Health Research Institute /ID# 145933, Washington D.C., District of Columbia
  - James A. Simon, MD, PC /ID# 139675, Washington D.C., District of Columbia
  - Helix Biomedics, LLC /ID# 147114, Boynton Beach, Florida
  - Brandon Premier Health Care, PA /ID# 153130, Brandon, Florida
  - Florida Clin Res Group /ID# 139811, Ckearwater, Florida
  - Universal Clinical Research A /ID# 139742, Doral, Florida
  - Clinical Physiology Associates /ID# 139736, Fort Myers, Florida
  - Meridien Research /ID# 139663, Kenneth City, Florida
  - Altus Research, Inc /ID# 139662, Lake Worth, Florida
  - South Florida Wellness & Clinic /ID# 143558, Margate, Florida
  - LCC Medical Research Institute /ID# 143551, Miami, Florida
  - Healthcare Clinical Data, Inc /ID# 139650, Miami, Florida
  - Ocean Blue Med Research Ctr /ID# 139826, Miami, Florida
  - Salom Tangir, LLC /ID# 151732, Miramar, Florida
  - Advanced Research Institute /ID# 143554, New Port Richey, Florida
  - Clinical Associates of Orlando /ID# 148123, Orlando, Florida
  - Omega Research Consultants /ID# 139648, Orlando, Florida
  - Unified Womens Clin Research /ID# 145169, Panama City, Florida
  - Comprehensive Clinical Trials /ID# 139644, West Palm Beach, Florida
  - Atlanta Medical Research Insti /ID# 147117, Alpharetta, Georgia
  - Paramount Research Solutions /ID# 139645, Alpharetta, Georgia
  - Agile Clinical Research Trials /ID# 143563, Atlanta, Georgia
  - Perimeter Inst Clinical Resear /ID# 148298, Atlanta, Georgia
  - Masters of Clinical Research, Inc. /ID# 139658, Augusta, Georgia
  - Fellows Research Alliance, Inc /ID# 139655, Savannah, Georgia
  - Boise Family Medical Center /ID# 139844, Boise, Idaho
  - Women's Health Practice, LLC /ID# 143569, Champaign, Illinois
  - Great Lakes Clinical Trials /ID# 148135, Chicago, Illinois
  - Affinity Clinical Research /ID# 150980, Oak Brook, Illinois
  - American Health Network of IN /ID# 139822, Avon, Indiana
  - GTC Research /ID# 141854, Kansas City, Kansas
  - Cypress Medical Research Ctr /ID# 147116, Wichita, Kansas
  - Research Integrity, LLC /ID# 139727, Owensboro, Kentucky
  - Clinical Trials Management, LLC - Covington /ID# 139651, Covington, Louisiana
  - Ochsner Baptist Medical Center /ID# 139740, New Orleans, Louisiana
  - Omni Fertility and Laser Insti /ID# 139836, Shreveport, Louisiana
  - Capital Women's Care /ID# 144109, Frederick, Maryland
  - Genesis Clinical Research - Fall River /ID# 148449, Fall River, Massachusetts
  - Great Lakes Research Group,Inc /ID# 139659, Bay City, Michigan
  - Grand Rapids Womens Health /ID# 139705, Grand Rapids, Michigan
  - Wayne State University Physician Group - Southfield /ID# 139802, Southfield, Michigan
  - Office of Edmond E. Pack, MD /ID# 139792, Las Vegas, Nevada
  - Mabey, Las Vegas, NV /ID# 148138, Las Vegas, Nevada
  - Lawrence OB/GYN /ID# 143567, Lawrenceville, New Jersey
  - Bosque Women's Care /ID# 145934, Albuquerque, New Mexico
  - Manhattan Medical Research /ID# 144471, New York, New York
  - Cwrwc /Id# 139664, Durham, North Carolina
  - Unified Women's Clinical Research-Greensboro /ID# 139829, Greensboro, North Carolina
  - Unified Women's Clinical Resea /ID# 139774, Raleigh, North Carolina
  - PMG Research of Wilmington LLC /ID# 152563, Wilmington, North Carolina
  - Unified Women's Clinical Resea /ID# 144721, Winston-Salem, North Carolina
  - University of Cincinnati /ID# 139820, Cincinnati, Ohio
  - Univ Hosp Cleveland /ID# 139741, Cleveland, Ohio
  - Complete Healthcare for Women /ID# 139673, Columbus, Ohio
  - Miami Valley Hospital /ID# 144430, Dayton, Ohio
  - University of Toledo /ID# 139787, Toledo, Ohio
  - Legacy Medical Group-Portland /ID# 148807, Portland, Oregon
  - Main Line Fertility Center /ID# 150295, Bryn Mawr, Pennsylvania
  - Penn State University and Milton S. Hershey Medical Center /ID# 139733, Hershey, Pennsylvania
  - Thomas Jefferson University /ID# 139812, Philadelphia, Pennsylvania
  - Temple University Hospital /ID# 151429, Philadelphia, Pennsylvania
  - Clinical Trials Research Svcs /ID# 139707, Pittsburgh, Pennsylvania
  - Medical University of South Carolina /ID# 148754, Charleston, South Carolina
  - Vista Clinical Research /ID# 139797, Columbia, South Carolina
  - WR-ClinSearch /ID# 143538, Chattanooga, Tennessee
  - Research Memphis Associates, LLC /ID# 139674, Memphis, Tennessee
  - Access Clinical Trials, Inc. /ID# 139730, Nashville, Tennessee
  - UT Southwestern Medical Center /ID# 143537, Dallas, Texas
  - Advances in Health, Inc. /ID# 139672, Houston, Texas
  - Victorium Clinical Research /ID# 149630, San Antonio, Texas
  - Discovery Clinical Trials-San Antonio /ID# 139776, San Antonio, Texas
  - Houston Ctr for Clin Research /ID# 149149, Sugar Land, Texas
  - Center of Reproductive Medicin /ID# 139813, Webster, Texas
  - Eastern Virginia Med School /ID# 139647, Norfolk, Virginia
  - Clinical Research Partners, LL /ID# 143999, North Chesterfield, Virginia
  - Clinical Trials Virginia, Inc. /ID# 139801, Richmond, Virginia
  - Emerson Clinical Research /ID# 147373, Vienna, Virginia
  - Seattle Women's Health, Research, Gynecology /ID# 139768, Seattle, Washington
  - Premier Clinical Research /ID# 148145, Spokane, Washington
  - Froedtert and Medical College /ID# 143566, Milwaukee, Wisconsin
- Canada (2):
  - IWK Health Center /ID# 149066, Halifax, Nova Scotia
  - The Ottawa Hospital /ID# 148695, Ottawa, Ontario
- Puerto Rico (2):
  - Rodriguez-Ginorio, San Juan /ID# 139847, San Juan
  - School of Medicine University of Puerto Rico-Medical Sciences Campus /ID# 139848, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Simon JA, Stewart EA, Jewell S, Li M, Snabes MC. Impact of demographic and clinical factors on elagolix plus add-back therapy effects on patient-reported nonbleeding symptoms in women with heavy menstrual bleeding and uterine fibroids: a post hoc analysis of data from two clinical trials. F S Rep. 2024 Jun 14;5(3):285-295. doi: 10.1016/j.xfre.2024.06.002. eCollection 2024 Sep. PMID 39381651
- [Derived] Beck D, Winzenborg I, Liu M, Degner J, Mostafa NM, Noertersheuser P, Shebley M. Population Pharmacokinetics of Elagolix in Combination with Low-Dose Estradiol/Norethindrone Acetate in Women with Uterine Fibroids. Clin Pharmacokinet. 2022 Apr;61(4):577-587. doi: 10.1007/s40262-021-01096-w. Epub 2021 Dec 8. PMID 34878624
- [Derived] Stewart EA, Archer DF, Owens CD, Barnhart KT, Bradley LD, Feinberg EC, Gillispie-Bell V, Imudia AN, Liu R, Kim JH, Al-Hendy A. Reduction of Heavy Menstrual Bleeding in Women Not Designated as Responders to Elagolix Plus Add Back Therapy for Uterine Fibroids. J Womens Health (Larchmt). 2022 May;31(5):698-705. doi: 10.1089/jwh.2021.0152. Epub 2021 Sep 28. PMID 34582715
- [Derived] Muneyyirci-Delale O, Archer DF, Owens CD, Barnhart KT, Bradley LD, Feinberg E, Gillispie V, Hurtado S, Kim JH, Wang A, Wang H, Stewart EA. Efficacy and safety of elagolix with add-back therapy in women with uterine fibroids and coexisting adenomyosis. F S Rep. 2021 May 26;2(3):338-346. doi: 10.1016/j.xfre.2021.05.004. eCollection 2021 Sep. PMID 34553161
- [Derived] Beck D, Winzenborg I, Gao W, Mostafa NM, Noertersheuser P, Chiuve SE, Owens C, Shebley M. Integrating real-world data and modeling to project changes in femoral neck bone mineral density and fracture risk in premenopausal women. Clin Transl Sci. 2021 Jul;14(4):1452-1463. doi: 10.1111/cts.13006. Epub 2021 Apr 8. PMID 33650259
- [Derived] Al-Hendy A, Bradley L, Owens CD, Wang H, Barnhart KT, Feinberg E, Schlaff WD, Puscheck EE, Wang A, Gillispie V, Hurtado S, Muneyyirci-Delale O, Archer DF, Carr BR, Simon JA, Stewart EA. Predictors of response for elagolix with add-back therapy in women with heavy menstrual bleeding associated with uterine fibroids. Am J Obstet Gynecol. 2021 Jan;224(1):72.e1-72.e50. doi: 10.1016/j.ajog.2020.07.032. Epub 2020 Jul 20. PMID 32702363
- [Derived] Schlaff WD, Ackerman RT, Al-Hendy A, Archer DF, Barnhart KT, Bradley LD, Carr BR, Feinberg EC, Hurtado SM, Kim J, Liu R, Mabey RG Jr, Owens CD, Poindexter A, Puscheck EE, Rodriguez-Ginorio H, Simon JA, Soliman AM, Stewart EA, Watts NB, Muneyyirci-Delale O. Elagolix for Heavy Menstrual Bleeding in Women with Uterine Fibroids. N Engl J Med. 2020 Jan 23;382(4):328-340. doi: 10.1056/NEJMoa1904351. PMID 31971678

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were randomized in a 1:1:2 ratio to 1 of 3 treatment groups: placebo, elagolix 300 mg BID, or elagolix 300 mg twice daily (BID) plus estradiol/norethindrone acetate (E2/NETA) once daily (QD).
Groups:
- Placebo: Placebo for both elagolix BID and E2/NETA QD
Period: Treatment Period
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Started (randomized) | 102 | 104 | 207
Randomized and Treated | 102 | 104 | 206
Completed (completed treatment period) | 83 | 81 | 164
Not Completed | 19 | 23 | 43
Period: Post-Treatment Follow-Up Period
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Started | 25 | 32 | 59
Completed | 17 | 24 | 29
Not Completed | 8 | 8 | 30
Not completed — Withdrawal by Subject | 2 | 6 | 7
Not completed — Lost to Follow-up | 3 | 0 | 13
Not completed — Required Surgery/Invasive Intervention | 2 | 2 | 2
Not completed — Other | 1 | 0 | 4
Not completed — Non-Compliance | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: All randomized and treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA | Total
Number analyzed (Participants) | 102 | 104 | 206 | 412
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (5.68) | 42.6 (5.16) | 42.6 (5.30) | 42.3 (5.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 104 | 206 | 412
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 4 | 34 | 57
  Not Hispanic or Latino | 83 | 100 | 172 | 355
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 1 | 2 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 70 | 69 | 141 | 280
  White | 30 | 27 | 59 | 116
  More than one race | 1 | 4 | 1 | 6
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting the Criteria for Responder
Description: Percentage of responders, defined as participants who met the following conditions:
  * Menstrual blood loss (MBL) volume < 80 mL during the Final Month (the last 28 days prior to and including the Reference Day, which is defined as the last visit date during the Treatment Period [last treatment visit date] or the last dose date if there are evaluable alkaline hematin data after the last treatment visit date and prior to or on the last dose date), and
  * ≥ 50% reduction in MBL volume from Baseline to the Final Month.
  Participants who prematurely discontinued study drug due to "lack of efficacy," "requires surgery or invasive intervention for treatment of uterine fibroids," or "adverse events" were considered non-responders regardless of whether she meets the two aforementioned responder criteria or not.
Time Frame: Final Month (the last 28 days prior to and including the Reference Day), up to Month 6
Population: All randomized and treated participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Number analyzed (Participants) | 102 | 104 | 206
percentage of participants | 8.7 | 84.1 | 68.5
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p < 0.001, Regression, Logistic — The P value for test of difference is by pooling the results from a logistic regression model including treatment as the main effect and baseline MBL volume as a covariate in each data set from multiple imputation; Odds Ratio (OR) = 56.79, 95% CI 2-sided [23.002 to 140.227]
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 22.98, 95% CI 2-sided [10.466 to 50.451]

2. Secondary Outcome: Change From Baseline in MBL Volume to the Final Month
Description: Baseline MBL volume was defined as the mean of total MBL volume from all the qualified menstrual cycles during the Screening Period, in which the total MBL volume is from all validated and non-validated sanitary products and the MBL volume of validated sanitary products only (excluding non-validated sanitary products) was greater than 80 mL.
  The Reference Day is defined as the last visit date during the Treatment Period (last treatment visit date) or the last dose date if there are evaluable alkaline hematin data after the last treatment visit date and prior to or on the last dose date.
Time Frame: Month 0 (Baseline), Final Month (the last 28 days prior to and including the Reference Day), up to Month 6
Population: All randomized and treated participants.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Number analyzed (Participants) | 102 | 104 | 206
mL | 0.8 (14.86) | -221.5 (14.49) | -176.7 (10.40)
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p < 0.001, ANCOVA — The P value for test of difference between each elagolix treatment group and placebo is by pooling the results from an ANCOVA model with treatment as the main effect and baseline MBL volume as a covariate in each dataset from multiple imputation; LS Mean of Difference = -222.3, Standard Error of Mean 20.77
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean of Difference = -177.5, Standard Error of Mean 18.24

3. Secondary Outcome: Percentage of Participants With Suppression of Bleeding at the Final Month
Description: Suppression of bleeding is defined as having 0 days of bleeding (spotting is allowed) during the Final Month with the interval starting from Study Day 11.
  The Reference Day is defined as the last visit date during the Treatment Period (last treatment visit date) or the last dose date if there are evaluable alkaline hematin data after the last treatment visit date and prior to or on the last dose date.
Time Frame: Final Month (the last 28 days prior to and including the Reference Day), up to Month 6
Population: All randomized and treated participants with an assessment
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Number analyzed (Participants) | 91 | 94 | 183
percentage of participants | 4.4 | 84.0 | 56.8
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p < 0.001, Chi-square or Fisher's exact test — The P value is calculated based on chi-square test (or Fisher's exact test if ≥ 20% of the cells have expected cell count < 5); Between-Group Difference (%) = 79.6, 95% CI 2-sided [71.13 to 88.16]
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Test type: Superiority; p < 0.001, Chi-square or Fisher's exact test — [p-value comment as in outcome 3, analysis 1]; Between-Group Difference (%) = 52.4, 95% CI 2-sided [44.11 to 60.76]

4. Secondary Outcome: Change From Baseline in MBL Volume to Month 6
Time Frame: Month 0 (Baseline), Month 6
Population: All randomized and treated participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Number analyzed (Participants) | 71 | 67 | 132
mL | -2.3 (13.53) | -236.2 (13.74) | -194.7 (9.77)
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p < 0.001, mixed model repeated measures — The P value is from mixed models repeated measures (MMRM) with treatment, month, and an interaction between treatment and month as fixed effect factors, and baseline MBL volume as a covariate comparing each elagolix treatment group with placebo; LS Mean of Difference = -234.0, Standard Error of Mean 19.27
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Test type: Superiority; p < 0.001, mixed model repeated measures — [p-value comment as in outcome 4, analysis 1]; LS Mean of Difference = -192.5, Standard Error of Mean 16.70

5. Secondary Outcome: Change From Baseline in MBL Volume to Month 3
Time Frame: Month 0 (Baseline), Month 3
Population: All randomized and treated participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Number analyzed (Participants) | 85 | 83 | 172
mL | 6.1 (15.32) | -234.7 (15.38) | -192.2 (10.81)
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p < 0.001, mixed model repeated measures — The P value is from MMRM with treatment, month, and an interaction between treatment and month as fixed effect factors, and baseline MBL volume as a covariate comparing each elagolix treatment group with placebo; LS Mean of Difference = -240.8, Standard Error of Mean 21.69
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Test type: Superiority; p < 0.001, mixed model repeated measures — [p-value comment as in outcome 5, analysis 1]; LS Mean of Difference = -198.2, Standard Error of Mean 18.76

6. Secondary Outcome: Percentage of Participants With Baseline Hemoglobin <= 10.5 g/dL Who Have an Increase in Hemoglobin > 2 g/dL at Month 6
Time Frame: Month 0 (Baseline), Month 6
Population: All randomized and treated participants with baseline hemoglobin <= 10.5 g/dL and an assessment at Month 6.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Number analyzed (Participants) | 31 | 41 | 52
percentage of participants | 16.1 | 65.9 | 61.5
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p < 0.001, chi-square or Fisher's exact test — [p-value comment as in outcome 3, analysis 1]; Between-Group Difference (%) = 49.7, 95% CI 2-sided [30.27 to 69.18]
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Test type: Superiority; p < 0.001, chi-square or Fisher's exact test — [p-value comment as in outcome 3, analysis 1]; Between-Group Difference (%) = 45.4, 95% CI 2-sided [26.90 to 63.92]

7. Secondary Outcome: Change From Baseline in MBL Volume to Month 1
Time Frame: Month 0 (Baseline), Month 1
Population: All randomized and treated participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: mL
Groups:
- Elagolix + Estradiol/Norethindrone Acetate: Elagolix 300 mg BID and E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) QD
Arm/Group | Placebo | Elagolix | Elagolix + Estradiol/Norethindrone Acetate
Number analyzed (Participants) | 95 | 97 | 187
mL | -19.0 (16.05) | -209.0 (15.91) | -135.2 (11.41)
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p < 0.001, mixed model repeated measures — [p-value comment as in outcome 5, analysis 1]; LS Mean of Difference = -190.0, Standard Error of Mean 22.59
Statistical Analysis 2: Comparison: Placebo vs Elagolix + Estradiol/Norethindrone Acetate; Test type: Superiority; p < 0.001, mixed model repeated measures — [p-value comment as in outcome 5, analysis 1]; LS Mean of Difference = -116.2, Standard Error of Mean 19.70

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 6 months of treatment with a 30-day follow-up period for participants who did not enroll in the extension study (Study M12-816). Mean (SD) treatment exposure was 158.6 (50.10), 161.2 (51.45), and 159.9 (53.48) days for the Placebo, Elagolix, and Elagolix and E2-NETA arms, respectively.
Description: Treatment-emergent adverse events are presented.
Groups:
- Elagolix + E2-NETA: Elagolix 300 mg BID and E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) QD
Arm/Group | Placebo | Elagolix | Elagolix + E2-NETA
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/104 | 0/206
Serious Adverse Events (participants affected / at risk) | 5/102 | 3/104 | 3/206
Other Adverse Events (participants affected / at risk) | 29/102 | 81/104 | 96/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=102) | Elagolix (N=104) | Elagolix + E2-NETA (N=206)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
PROLAPSE (General disorders) | 0 (0) | 1 (1) | 0 (0)
OXYGEN SATURATION DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PALMOPLANTAR KERATODERMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=102) | Elagolix (N=104) | Elagolix + E2-NETA (N=206)
NAUSEA (Gastrointestinal disorders) | 10 (10) | 7 (7) | 23 (26)
FATIGUE (General disorders) | 2 (2) | 1 (1) | 14 (14)
NASOPHARYNGITIS (Infections and infestations) | 4 (5) | 6 (6) | 10 (12)
HEADACHE (Nervous system disorders) | 9 (11) | 17 (20) | 17 (18)
INSOMNIA (Psychiatric disorders) | 6 (6) | 7 (7) | 5 (5)
MOOD SWINGS (Psychiatric disorders) | 2 (2) | 7 (7) | 8 (8)
DYSMENORRHOEA (Reproductive system and breast disorders) | 4 (4) | 1 (1) | 13 (13)
METRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 13 (13)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 3 (3) | 28 (31) | 14 (15)
HOT FLUSH (Vascular disorders) | 9 (10) | 67 (72) | 42 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT02654054/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT02654054/SAP_001.pdf